CLINICAL TRIAL: NCT06349720
Title: A Study of the Trajectory of Overall Systemic Health Outcomes and Potential Complications in Recovered COVID-19 Patients.
Brief Title: Investigating Long-term Health Effects and Complications in COVID-19 Recoveries
Status: Recruiting | Type: Observational
Sponsor: Zhaohui Tong (Other)
Responsible Party: Sponsor-Investigator, Zhaohui Tong, professor, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: KF-2023-355
Record Dates: First submitted 2024-04-03; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- severe vs non-severe
- COVID-19 patients vs healthy volunteers
- emote respiratory rehabilitation vs outpatient respiratory rehabilitation
  Interventions: Behavioral: respiratory rehabilitation

INTERVENTIONS:
Behavioral: respiratory rehabilitation — Emote respiratory rehabilitation:Patients wear monitoring devices and upload real-time monitoring data such as vital signs through the FREE rehabilitation app installed on their personal phones. Medical staff monitor changes in patients' vital signs in real time through the FREE rehabilitation app on the medical end, and adjust respiratory rehabilitation plans based on their phone or video guidance.
  Outpatient respiratory rehabilitation:Traditional outpatient respiratory rehabilitation is based on a group approach, with individualized intensity determined based on baseline assessment results, and is conducted under supervision twice a week for a period of 12 weeks.
  Groups: emote respiratory rehabilitation vs outpatient respiratory rehabilitation

SUMMARY:
Clarify the incidence of functional impairments in cured COVID-19 patients and identify influencing factors. Build a multi-omics database for COVID-19 patients in the recovery period to elucidate the biological biomarkers and targets associated with functional impairments. Comprehensive exploration of the long-term prognosis, complications, sequelae, and risk factors of COVID-19 patients after Omicron infection, as well as their immune characteristics. Compare the impact of different strains of the COVID-19 virus on prognosis and immune response. Develop comprehensive rehabilitation intervention strategies for COVID-19 patients with functional impairments and evaluate the impact of different intervention methods on their prognosis. Based on clinical data, multi-omics data, and precise rehabilitation assessment data, construct predictive models for prognosis and rehabilitation effectiveness in COVID-19, providing scientific evidence for the implementation of effective COVID-19 rehabilitation measures.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for confirmed cases according to the "Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 10)";
2. The participant or the authorized representative understands the entire purpose of the study, voluntarily participates in the research, and signs an informed consent form, ensuring that they can complete regular assessments at the relevant participating units and receive necessary rehabilitation treatment as required;
3. Agrees to the researcher's collection of their peripheral blood samples, saliva samples, and urine samples for the needs of the study.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. Individuals with mental disorders that affect normal communication;
3. Those who refuse to participate in regular assessments and rehabilitation treatments;
4. Individuals who decline to provide specimens required for the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital
Sampling Method: Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Immunological characteristics associated with functional impairments in COVID-19 convalescent patients | 6 months, 12 months and 24 months
Changes in laboratory examination indicators | 6 months, 12 months and 24 months
High-resolution CT of the chest | 6 months, 12 months and 24 months
Pulmonary function test | 3 months, 12 months
Multi-omics changes and characteristics associated with functional impairments in COVID-19 convalescent patients | 6 months, 12 months and 24 months
Inflammatory factors related to body dysfunction in COVID-19 rehabilitation patients | 6 months, 12 months and 24 months
Regular rehabilitation assessment following respiratory rehabilitation intervention in COVID-19 patients | 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes